CLINICAL TRIAL: NCT03157245
Title: Interest of Doppler Ultrasound for the Assessment of Incidence of Deep Vein Thrombosis on Central Venous Catheters in the Post Operative Period of Carcinologic Surgery
Brief Title: Incidence of Deep Vein Thrombosis on Central Venous Catheters in the Post Operative Period of Carcinologic Surgery
Acronym: THROMBOCAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A00043-50
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Critically Ill; Central Venous Catheter Thrombosis; PARENTERAL NUTRITION; POST OPERATIVE
MeSH Terms: conditions — Critical Illness; Upper Extremity Deep Vein Thrombosis; Hyperphagia | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- participant
  Interventions: Diagnostic Test: DOPPLER ULTRASOUND

INTERVENTIONS:
Diagnostic Test: DOPPLER ULTRASOUND — MESURE OF THE PRESENCE OR NOT OF A CATHETER RELATED VEIN THROMBOSIS

SUMMARY:
The objective is to determine the incidence of thrombosis on central venous catheters in patients hospitalized in a surgical critical care unit, in the immediate postoperative period of urological or digestive carcinological surgery, and receiving parenteral nutrition.

DETAILED DESCRIPTION:
The post operative period, wich is a critically ill condition, and history of cancer are related to a high risk of venous thrombosis. Catheter is one of the most common complication of parenteral nutrition and is also related to thrombosis.

The combination of theses conditions increases the risk of venous catheter thrombosis. , Since, there is no data evaluating this risk nowadays, the objective of this study is to determine the incidence of thrombosis on central venous catheters in patients hospitalized in a surgical critical care unit, in the immediate postoperative period of urological or digestive carcinological surgery, and receiving parenteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in surgical intensive care in the immediate post-operative period
* surgery for cancer
* central venous catheter placement for parenteral nutrition
* written consent dated and signed before doppler examination

Exclusion Criteria:

* patient < 18 years old
* pregnancy
* surgery with no indication for parenteral nutrition on central venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient > 18 years old, admitted in surgical critical care, immediatly after elective carcinologic surgery with a central venous catheter for parenteral nutrition
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Presence or no of a catheter related thrombosis | 1 day (day of the catheter removal)
  Patients will undergo an examination by a specialist in vascular medicine just before removal of the catheter.This specialist also is specialist in vascular doppler ultrasonography.
  The specialist would search symptoms and signs of deep vein thrombosis : local pain, swelling, redness, warmth. Clinical examinated would be completed by doppler ultrasound : thrombus is detected during a compression test, while cruor is evaluated in B-mode (gray-scale) imaging. This method is very sensitive with regard to detection of the thrombus.

SECONDARY OUTCOMES:
clinical factors associated with the presence of catheter related thrombosis | post operative period, during the intensive care unit stay
  During the intensive care unit stay, the investigator would prospectively collected data, including :
  * potential risk factors : age, history of venous thrombosis, type of cancer...
  * details of surgery : type and operating time
  * details of critically ill period : number and type of organs failures, first mobilisation..
  * details of the clinical course : occurence of a situation requiring curative anticoagulation..

CONTACTS AND LOCATIONS:
Locations (1):
- NOVY, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No